CLINICAL TRIAL: NCT06698328
Title: Developing Brain Imaging Biomarkers to Quantify the Effects of At-home taVNS Treatment in ASD
Brief Title: fMRI Tracking taVNS in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC COBRE in Neurodevelopment and its Disorders (CNDD) Pilot Projects Program (PPP) (Unknown)
Responsible Party: Principal Investigator, Xiaolong Peng, Research Instructor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00140411
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autistic Spectrum Disorders
Keywords: Adolescents; Anxiety; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Vagus Nerve Stimulation (Active Comparator): This active vagus nerve stimulation uses electrodes on the ear to be administered twice daily, seven days per week, for four weeks at-home.
  Interventions: Device: Transauricular Vagus Nerve Stimulation
- Sham Stimulation (Sham Comparator): This sham nerve stimulation uses electrodes on the ear to be administered twice daily, seven days per week, for four weeks at-home.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transauricular Vagus Nerve Stimulation — Mild non-invasive electrical stimulation to the vagus nerve using electrodes or "stickers" that adhere to the ear and the surrounding area.
  Arms: Active Vagus Nerve Stimulation
Device: Sham Stimulation — Sham non-invasive electrical stimulation using electrodes or "stickers" that adhere to the ear and the surrounding area.
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to explore whether a non-invasive form of ear stimulation called transcutaneous auricular vagus nerve stimulation (taVNS) can manage symptoms in patients with autism spectrum disorder (ASD). Additionally, this study also uses magnetic resonance imaging (MRI) to capture images of participants' brains and apply an image processing method called INSCAPE to track brain state changes during taVNS treatment in ASD. Investigators will recruit up to 16 participants with ASD.

DETAILED DESCRIPTION:
In this study, the Investigators main goal is to establish and validate new imaging biomarkers for evaluating and tracking changes in functional networks and dynamic brain states that occur over 1-month transcutaneous auricular vagus nerve stimulation (taVNS) treatment in individuals with autism spectrum disorder (ASD) at home.

In this double-blinded sham-controlled clinical trial, Investigators will recruit up to 16 patients with ASD and co-occurring anxiety symptoms from the outpatient clinics at MUSC, SPARK, Epic, and social media (i.e., Project Rex, SCARO). Each participant will first receive the baseline behavior evaluation using a neuropsychiatric battery. Then, participants will have a high-resolution structural MRI scan and four runs of resting-state fMRI scans (~30-min in total) at MUSC 30 Bee Street Center for Biomedical Imaging. This will be followed by an in-person training session with the subject (and legal guardian if applicable), where they will learn how to self-administer taVNS and ask any pertinent questions. Participants will self-administer taVNS (or sham) at home twice daily for 4 weeks. At the end of 4 weeks, participants will have the post-taVNS MRI scanning and behavioral evaluation. Additionally, participants will also complete the behavioral evaluation virtually right after the 2-week treatment, and follow-up 1 and 4 weeks after the completion of treatment.

Aim 1. Identify dynamic imaging biomarkers capable of tracking the brain state changes of ASD throughout a one-month taVNS treatment at home.

Aim 2. Explore whether dynamic brain state measures derived from baseline can predict symptom improvement and response to taVNS treatment.

Results from this study may help to further optimize this taVNS therapy and lead to more effective treatment for ASD, as well as identify dynamic imaging biomarkers that can quantify and track symptom recovery in this unique population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-17
* English speaking
* Prior diagnosis of ASD using autism diagnostic observation schedule (ADOS)
* Have the capacity and ability to provide one's own assent, consent will be provided by legal guardian

Exclusion Criteria:

* Facial/ear pain or recent ear trauma
* Metal implant devices in the head, heart, or neck
* History of brain surgery
* History of myocardial infarction or arrhythmia/bradycardia
* Acute exacerbation of a chronic respiratory disorder or acute COVID-related symptoms
* Active GI symptoms with a history of diabetes mellitus (DM) or gastroparesis secondary to DM
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium)
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury
* Personal history of frequent/severe headaches
* Personal history of psychosis or mania, or individuals who are actively manic or psychotic
* Individuals who are catatonic or otherwise unable to participate in the informed consent process
* Moderate to severe alcohol or substance use disorder
* Pregnancy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing adverse outcomes as measured by questionnaire | 1 month of experimental at-home taVNS treatment
  Assessing adverse outcomes via qualitative questionnaire asking participants about experiences during stimulation and any consequences after stimulation.

SECONDARY OUTCOMES:
Dynamic Brain States Change Relative to ASD through fMRI | fMRI imaging will be conducted at baseline and at the 1 month follow-up final visit
  Participants will undergo two MRI scans looking at the changes in brain states. One scan will be prior to stimulation treatment and one scan will be after one month of stimulation treatment.
Anxiety rating for participants using the generalized anxiety disorder -child scale | Through study completion, up to 2 months
  Assessing the impact of stimulation on GAD-child scale, where lower numbers (0=none, 4=extreme) show improved anxiety
Empagthic abilities as measured by the Toronto Empathy Questionnaire | Through study completion, up to 2 months
  Assessing the participants change in the ability to identify the emotions of others using the TEQ, while a score of less than 45 indicating below average empathy levels, and a max score of 64

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Peng, Principal Investigator — Medical University of South Carolina
Locations (1):
- 30 Bee Street, Charleston, South Carolina, United States